CLINICAL TRIAL: NCT03639298
Title: Premature Children-executive Functions and Training With Cognitive Motion-based Videogames (Intendu®): a Rehabilitation Project
Brief Title: Executive Functions Rehabilitation in Premature Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to SARS-Cov-2 emergency we were unable to recruit the expected number of children. We will analyze the available data
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Barbara Scelsa, MD, Vittore Buzzi Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BS1
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Executive Functions
Keywords: premature children; processing speed; executive functions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training (Experimental): children submitted to the Intendu training with motion based cognitive video games software
  Interventions: Device: Intendu
- no training (No Intervention): children not submitted to the training, entering the study as a control group

INTERVENTIONS:
Device: Intendu — intensive training with Motion Based Cognitive Video Games Software
  Arms: training

SUMMARY:
in more than 60% of premature children processing speed and academic failures are observed, even in children with a normal cognitive level.

The aim of the study is to use for rehabilitation an application for training functional cognitive skills (Intendu®). It is a software which is able to interact with the patient through a video monitoring feedback (Kinect®), enhancing brain plasticity of patients with brain dysfunction.

DETAILED DESCRIPTION:
In Europe 6.2% of the births are born before 37 weeks of gestation. After a long period in Neonatal Intensive Care Units, the infants are dismissed but they continue to be examined in follow-up programs. It is known that advances in care have improved the rate of survival of premature newborns, but unfortunately they may have disabilities which can be severe (cerebral palsy) or mild. Mild disabilities (like attention deficit, hyperactivity, visual-perceptual and coordination disorders), even if mild, can have a significant impact on school achievements and social life. Follow-up program is dedicated to detect both severe and minor disabilities, trying to rehabilitate the children before they start formal education in school. It is well known that more than half of premature children can show impairment of processing speed and academic failures, even with normal cognitive level. Processing speed is the result of the action of different executive functions, especially working memory, planning, attention shift, inhibition and persistence.

There is growing interest over cognitive rehabilitation with video games. Recently an application for training functional cognitive skills (Intendu®) has been developed . It is a software which is able to interact with patients through a video monitoring feedback (Kinect®), enhancing brain plasticity of patients with brain dysfunction.

Aim of the study:

To evaluate whether an adaptive motion-interaction video game can improve processing speed and executive functions in premature children.

Methods:

35 children born prematurely (23-36.5 W) aged 4-6 year-old with reduced processing speed, will be invited to participate if they meet the inclusion criteria. They will be submitted to 4-5 weeks intensive training with Intendu®, (4-5 sessions per week, for a total of 20 sessions) lasting 15 minutes each, in the presence of a tutor (a psychologist expert in premature children). A control group of 35 children (no training) with the same characteristics (gestational age, cognitive profile, socio-economic status) will be available. Before and after the training/or no training the participants, in addition to the scheduled follow-up assessment, will be evaluated with two WPPSI-III®-Wechsler Preschool and Primary Scale of Intelligence subtests (Coding and Symbol search) and one Nepsy II® domain-A developmental Neuropsychological Assessment (attention and executive function). Teacher and parents evaluations will be also considered (school reports and Child Behavior Checklist - questionnaire)

ELIGIBILITY:
Inclusion Criteria: children

* born between 23-36.5 weeks of gestation
* age between 4 and 0 month -6 years and 11 months
* included in the V, Buzzi children's Hospital follow-up program
* resident no further than 20 km from the V. Buzzi Children's Hospital
* with WPPSI-III processing speed quotient of 91 or less

Exclusion Criteria:

* children affected by epilepsy

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
change in WPPSI-III ( Wechsler Preschool and Primary Scale of Intelligence) Processing Speed Quotient | assessment at baseline (time 0) and at the end of the training (after 4 weeks)
  the achievement of at least 10 points change of WPPSI® Processing Speed Quotient (subtests: Coding and Symbol search) will be considered significant
change in scaled scores of Nepsy II® (developmental Neuropsychological Assessment) attention and executive function domain | assessment at baseline (time 0) and at the end of the training (after 4 weeks)
  the achievement of at least 3 points change in scaled scores of Nepsy II® attention and executive function domain

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Scelsa, MD, Principal Investigator — V. Buzzi Children's Hospital
Locations (1):
- V. Buzzi Children's Hospital, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No
protocol of the study and patient data

REFERENCES:
- [Background] Volpe JJ. Brain injury in premature infants: a complex amalgam of destructive and developmental disturbances. Lancet Neurol. 2009 Jan;8(1):110-24. doi: 10.1016/S1474-4422(08)70294-1. PMID 19081519
- [Background] Johnson S. Cognitive and behavioural outcomes following very preterm birth. Semin Fetal Neonatal Med. 2007 Oct;12(5):363-73. doi: 10.1016/j.siny.2007.05.004. Epub 2007 Jul 10. PMID 17625996
- [Background] Dye MW, Green CS, Bavelier D. Increasing Speed of Processing With Action Video Games. Curr Dir Psychol Sci. 2009;18(6):321-326. doi: 10.1111/j.1467-8721.2009.01660.x. PMID 20485453